CLINICAL TRIAL: NCT05567432
Title: Hemostasis in Thyroidectomy, Comparison Between Diathermy and Ligasure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Aboelhassan Guishy, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: htdl
Record Dates: First submitted 2022-09-17; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Thyroid
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroidectomy

STUDY DESIGN:
Intervention Model Description: In about 20 participants , the investigators will control bleeding and cut tissues and blood vessels using the diathermy and in the other 20 , investigators will do homeostasis with ligasure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will do throidectomy using diathermy (Active Comparator): In these patients the investigators will control bleeding and cut tissues and blood vessels using the diathermy .
  Interventions: Procedure: thyroidectomy
- Patients will do thyroidectomy using ligasure . (Active Comparator): In these patients the investigators will control bleeding and cut tissues and blood vessels using the liagasure.
  Interventions: Procedure: thyroidectomy

INTERVENTIONS:
Procedure: thyroidectomy — use diathermy or ligasure for homeostatic during thyroidectomy

SUMMARY:
Thyroidectomy is one of the most surgeries done by surgeons. Postoperative bleeding is a main complication for this surgery.surgeons usually do homeostasis by traditional diathermy as it is cheep and available in all hospitals and centres.

Atlternatinve surgery devices have become popular to conventional hemostasis in thyroid surgery. These devices reduce operative time and post-operative complication .Investigators thought to examine relative efficiency of two alternative energy devices compared to each other in preventing post-operative complication between diathermy and ligasure.

DETAILED DESCRIPTION:
Thyroid surgery is one of the most frequently performed surgical procedures worldwide . Nowadays, total thyroidectomy is the recommended procedure for thyroid disease . As total thyroidectomy is the procedure of choice, the most common complication resulting after this surgery is transient hypocalcemia - the incidence being 24% - which increases the morbidity rate and increases the length of hospitalization. Other complications of thyroidectomy include recurrent laryngeal nerve injury which leads to hoarseness of voice, postoperative hemorrhage, dysphagia due to inflammation of the tissues surrounding the esophagus, seroma formation, Horner's syndrome due to injury to the cervical sympathetic chain, and poor healing of the wound with hypertrophy of the scar or wound infection .

Atlternatinve surgery devices have become popular to conventional hemostasis in thyroid surgery. These devices reduce operative time and post-operative complication .Investigators thought to examine relative efficiency of two alternative energy devices compared to each other in preventing post-operative complication between diathermy and ligasure.

ELIGIBILITY:
Inclusion Criteria:

* • Patient with disburbed thyroid function and candidate for for thyroidectomy

Exclusion Criteria:

* Low preoperative calcium level and Patient with contraindication of uses of ligasure or diathermy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Finding the best methode to decrease intraoperative and postoperative bleeding during thyroidectomy | 6 months
  This study is aiming to make a comparison between the incidence of intraoperative and postoperative bleeding while using diathermy versus using ligasure in homeostasis during thyroidectomy.
  * The investigators will do their best to answer this question... 1. ls rate of postoperative complications decrease while using the ligasure than using traditional diathermy ?

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Korany, PHD, Study Director — Assut University

REFERENCES:
- [Background] Manouras A, Markogiannakis H, Koutras AS, Antonakis PT, Drimousis P, Lagoudianakis EE, Kekis P, Genetzakis M, Koutsoumanis K, Bramis I. Thyroid surgery: comparison between the electrothermal bipolar vessel sealing system, harmonic scalpel, and classic suture ligation. Am J Surg. 2008 Jan;195(1):48-52. doi: 10.1016/j.amjsurg.2007.01.037. PMID 18082542